CLINICAL TRIAL: NCT05481164
Title: Population-based New-Born Screening of Spinal Muscular Atrophy to Evaluate the Uptake and Feasibility in the UK Context
Brief Title: Newborn Screening for Spinal Muscular Atrophy
Acronym: SMA-NBS
Status: Completed | Type: Observational
Sponsor: University of Oxford (Other)
Collaborators: Novartis Gene Therapies (Industry); Hoffmann-La Roche (Industry); Oxford University Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: Oxford
Record Dates: First submitted 2022-06-21; First posted 2022-08-01 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-09

CONDITIONS: Muscular Atrophy, Spinal
MeSH Terms: conditions — Muscular Atrophy, Spinal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — an automated multi-hole punching machine generates samples (discs) from the dried blood spots on the Guthrie card, to be used in the routine screening of conditions included in national NHS newborn blood spot screening programme.
  DNA will be extracted from the sample and run on a sensitive assay called qPCR, which will allow us to detect the presence of the affected gene in SMA, called SMN1.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Screen for Spinal Muscular atrophy for newborns: Babies with an SMA screen-positive result

SUMMARY:
Spinal muscular atrophy (SMA) is a rare, treatable, genetic disease that typically occurs in infancy and early childhood. SMA progressively, and irreversibly, destroys motor neurons in the brainstem and spinal cord, which control movement, in turn leading to deterioration or loss of muscle strength.

This can begin during the first 3 months of a child's life, and in those with the most common and severe type of SMA, 95% of all motor neurons can be lost before the age of 6 months. The majority of children with this type of SMA, if untreated, will not survive beyond 2 years of age without permanent ventilatory support. Of those who do, many will not achieve independent sitting and few walk independently.

A challenging aspect of treating SMA is the delay in its diagnosis, usually after disease onset. Diagnosis usually occurs when the affected child presents clinical symptoms, by which point a significant portion of their motor neurons will have been irreversibly lost. In contrast, infants and children with SMA who are identified and treated at an early stage, especially those treated pre-symptomatically, show much better motor development.

Given that SMA is caused by deletions or mutations in the survival motor neuron 1 gene (SMN1), it can be detected via genetic testing before a child presents with clinical symptoms. This lends itself to newborn genetic screening, through which pre-symptomatic diagnosis of SMA can be made as early as possible, providing the opportunity for substantially enhanced therapeutic effects and outcomes.

The aim and objective of this screening study is to assess the uptake, reliability, and feasibility of neonatal screening for SMA in a UK setting. It is hoped that by doing so it will help establish the early detection, diagnosis, and access to the recently available therapeutic options for SMA.Screening will be done through the routine UK newborn blood spot screening pathway, using spare capacity from a newborns' Guthrie card (dried blood spot sample). A major objective of the design of this protocol and the processes it describes, together with the staff funding secured, has been to ensure that it will not interfere with the standard screening procedure in any way.Recruitment will be carried out in the maternity units of four hospital trusts in the Thames Valley: Oxford University Hospitals NHS Trust, Royal Berkshire NHS Foundation Trust, Milton Keynes University Hospital NHS Foundation Trust, and Buckinghamshire Healthcare NHS Trust.

DETAILED DESCRIPTION:
Spinal muscular atrophy (SMA) is a progressive, debilitating neuromuscular disorder that leads to the deterioration or loss of muscle strength, including that of the respiratory muscles, and continues to be the most common inheritable cause of infant mortality. SMA affects about 1/10,000 newborns. Although the age at symptom onset may vary, it most frequently occurs in infancy and early childhood, with more severe clinical phenotypes correlating with earlier symptom onset. In Type 1 SMA, which is both the most common and severe form of the disease, symptom onset typically occurs by the age 6 months. A majority of these patients, if untreated, will not survive beyond 2 years of age in the absence of permanent ventilation support; of those who do, many will not achieve independent sitting, and few, if any, will walk independently. In the relatively milder but less common Types 2 and 3 SMA, patients have a lower or largely normal lifespan but, if untreated, still frequently lose ambulation over time, even when it had previously been acquired. These clinical phenotypes, resulting from the loss of motor function, are driven by the irreversible degeneration and loss of motor neurons in the spinal cord. This begins during the first 3 months of life and, in patients with Type 1 SMA, 95% are lost before the age of 6 months. As a result , a significant portion of motor neurons may be irreversibly lost before symptoms appear, and before a clinical diagnosis can be made. Given this, a screening method that would facilitate earlier diagnosis and hence treatment, before pathophysiological deterioration, is necessary.

SMA is caused by deletions or mutations in the survival motor neuron 1 (SMN1) gene, which can be detected through genetic testing before patients present clinical symptoms. This lends itself to newborn genetic screening, through which pre-symptomatic diagnosis of SMA patients can be made as early as possible, providing the opportunity for better therapeutic effects. As a genetic diagnosis, qPCR or MLPA present a 100% specificity, and a 100% sensitivity for the homozygous deletion. For patients with an heterozygous deletion and a point mutation, the diagnosis is done by qPCR and gene sequencing. In the current study, we will use qPCR as a first tier diagnosis.

There are currently three treatments available to SMA patients that can significantly improve their prognosis, particularly with early intervention. All of these treatment methods have shown to be able to target the underlying genetic cause of SMA, as opposed to providing palliative and symptomatic care. Nusinersen, approved by the European Medicines Agency (EMA) in June 2017 and reimbursed by The National Institute for Health and Care Excellence (NICE) since June 2019, is an antisense oligonucleotide treatment that is administered intrathecally to modify the gene splicing of the 'back-up' SMN2 gene, compensating for the reduced levels of SMN proteins in patients with SMA. Risdiplam, which shares a similar mechanism of action to Nusinersen, is an orally-available treatment, and is currently under review for approval by the EMA. Zolgensma, approved by the EMA in March 2020 and currently under review for reimbursement by NICE, is a one-time gene therapy, delivered in a single intravenous dose, that replaces the impaired SMN gene in patients with SMA.

While treatment efficacy has been established in the clinical trial studies for these therapeutic options, patient age and time from symptom onset to the start of treatment have been identified as predictive factors of treatment efficacy options. In two early Nusinersen trials with symptomatic patients (ENDEAR: NCT02193074 and CHERISH: NCT02292537), the treatment was found to be more effective when administered early. In ENDEAR, which focused on the treatment of early-onset patients, subgroup analyses showed that those who received Nusinersen treatment earlier in their disease course demonstrated an increased likelihood of both event-free survival and motor development improvement from baseline assessment. Similarly, CHERISH, which focused instead on the treatment of later-onset patients, observed greater improvements in motor function assessments from baseline among those with shorter disease duration at screening. The ongoing Risdiplam trials with symptomatic patients (FIREFISH: NCT02913482 and SUNFISH: NCT02908685) have corroborated this observation. In FIREFISH, early-onset patients (SMA1) treated with Risdiplam sooner in their disease course showed greater improvement in motor function, with the same also observed in SUNFISH with later-onset patients (SMA2 and 3). A Zolgensma trial for post-symptomatic SMA1 patients (START: NCT02122952) further showed that, regardless of a patient's initial disease severity (as measured by their baseline motor function), earlier treatment of the disease can lead to more significant motor function gains: Subgroup analysis revealed that patients who received Zolgensma treatment earlier into their disease progression showed a greater improvement in motor function when compared to those who received treatment later into their disease progression, despite the higher baseline motor function score of the latter group. Taken together, these studies point to the role of early intervention in yielding better clinical outcomes, irrespective of the treatment administered.

Building on this, more recent clinical trials with these treatment options have focused on identifying and treating patients pre-symptomatically. In the Nusinersen trial NURTURE (NCT02386553), which enrolled patients (≤42 days) who were pre-symptomatic with SMA, 88% acquired autonomous ambulation, and 100% survived without permanent ventilation; in an earlier trial ENDEAR (NCT02193074), which enrolled patients who were postsymptomatic with SMA, 0% acquired autonomous ambulation, and 61% survived without permanent ventilation. Data from a Zolgensma trial SPR1NT (NCT03505099), which similarly enrolled patients (≤42 days) who were pre-symptomatic with SMA, have also emphasised the value of early treatment. Since treatment initiation following early genetic diagnosis, SPR1NT patients have shown greater improvements in clinical motor assessments (CHOP-INTEND) in comparison with those enrolled and treated post-symptomatically in Zolgensma's earlier trial, START (NCT02122952). Furthermore, no SPR1NT patients have required ventilatory support, and all have shown age-appropriate motor development since pre-symptomatic treatment initiation. This never happens in post-symptomatic patients. A Risdiplam trial, RAINBOWFISH (NCT03779334), enrolling genetically diagnosed, pre-symptomatic patients (≤42 days), is also currently underway. Collectively, these studies emphasise the importance of early diagnosis of SMA, a key step to facilitating pre-symptomatic treatment.

Pre-clinical diagnosis via Newborn Screening SMA is typically detected and diagnosed clinically, often long after disease progression, and only with the onset of symptoms. To overcome these diagnostic delays that routinely place patients outside the most effective treatment windows, molecular genetic testing must be relied upon for SMA diagnosis. Globally, newborn genetic screening programmes for SMA have increased population access to timely diagnosis, and treatment of SMA. These timelines align with the most efficacious treatment windows, emphasising the effectiveness of using this public health tool in the pre-symptomatic diagnosis and treatment of SMA. This rationale has provided the impetus for several SMA newborn screening studies in Australia, Italy, Germany and Southern Belgium, as well as official programmes in 31 states in the USA, The Netherlands and Taiwan. These studies have, collectively, demonstrated the uptake and feasibility of population-based newborn screening for SMA. Studies have reported a >99% acceptability rate (approached mothers consenting to participate) with an opt-in strategy, and 100% with an opt-out strategy; One study recorded a 93.03% acceptability rate across three hospital sites even before the availability of a currently approved treatment. These studies have also demonstrated the feasibility of newborn genetic screening processes to reliably identify newborns who will develop SMA, reporting specificity rates (proportion of correct negative diagnoses) of 100% in Belgium, 100% in Taiwan, and 100% in New York state.

Molecular genetic tools to diagnose SMA are well established, and newborn bloodspot screening, an internationally established public health measure, is routinely carried out in the UK to detect newborns affected by congenital diseases. Given these points, and with prior studies showing the acceptability and feasibility of newborn screening processes for SMA elsewhere globally, these considerations collectively provide strong rationale for evaluating similar study endpoints for the newborn genetic screening of SMA in a pilot within the United Kingdom. Importantly, this study has been designed, as a first priority, to establish its ability to be undertaken without disturbing the official Newborn Screening (NBS) programme.

STUDY DESIGN This is a prospective, observational, population screening study designed to evaluate the uptake, reliability, and feasibility of newborn screening for SMA in a UK NBS pathway in the Thames Valley, with the goal of facilitating early diagnosis and treatment of SMA. This study will enrol newborns whose mother is in her second or third trimester of pregnancy (≥18 weeks' gestation), and up until they are 28 days post-natal.

As part of the standard, NHS newborn blood spot screening programme, newborns are routinely tested for nine treatable metabolic and hormonal disorders. For these tests, a few drops of blood, collected from a newborn's vein or heel, are collected onto specimen collection paper (the Guthrie card), normally within a week of birth. For newborns in this study, testing of their samples will be undertaken and processed at the Oxford Neonatal Screening Laboratory at the Oxford University Hospitals NHS Trust (which provides sample processing for all neonatal and antenatal screening in the Thames Valley). Specific consent provided by their mothers will allow the use of their residual blood spot samples for their genetic screening of SMA. No additional blood samples will be required.

The sample processing method will require no study-specific sampling, and no additional sampling from the newborn beyond the standard neonatal blood collection procedure performed for the national NHS newborn blood spot screening programme. Since the newborn would be enrolled into the study before this blood sampling procedure, the sample generated from this routine procedure will be used. In accordance with normal practice, their dried blood spot (Guthrie card) sample will be delivered to the Oxford Neonatal Screening Laboratory at the John Radcliffe Hospital, where an automated instrument will 'punch' out small discs from the dried blood spots for use in a range of routine tests for the national NHS newborn blood spot screening programme. For newborns following this processing protocol, the only additional step undertaken for this study, beyond routine practice, is the 'punching' of an additional disc from spare capacity on the card for the subsequent genetic testing for SMA. This study sample will subsequently be delivered to the NHS Oxford Regional Genetics Laboratories at the Churchill Hospital for DNA extraction and genetic testing.

ELIGIBILITY:
Inclusion Criteria:

* Whose mother is undergoing antenatal care at one of the four Hospital Trusts in the Thames Valley region, whose blood spot will be screened at the NHS Oxford Regenial Genetics Laboratory
* Whose mother is able to understand the participant information sheet and is willing to provide her informed consent.
* Whose mother is in the second or third trimester of pregnancy (≥18 weeks' gestation), or up to 28 days postnatal (the latter is consistent with the World Health Organisation's definition of a newborn infant or neonate)

Exclusion Criteria:

* Whose mother is unable to understand written or verbal English which would preclude them from understanding the study

Min Age: 16 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Women who are pregnant.
Study Population: Pregnant women
Sampling Method: Probability Sample
Enrollment: 33568 (Actual)
Dates: Start 2022-03-08 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
To assess the uptake of newborn bloodspot genetic screening for spinal muscular atrophy among expectant and delivered mothers over the course of the 36 month study | All outcome measures will be assessed intermittently over the course of the 36 month period of the study
  1. The number of approached mothers
  2. The number of consented mothers
  3. The proportion of approached mothers consenting to take part in the study, measured by the number of consented mothers divided by the combined total of consented and approached mothers (times 100%)
  4. The number of SMA samples processed at the NHS neonatal and antenatal Screening Laboratory at the John Radcliffe Hospital

SECONDARY OUTCOMES:
To determine the feasibility and reliability of the study screening test and regimen in identifying true positive cases | All outcome measures will be assessed intermittently over the course of the 36 month period of the study
  1. The number of false positive results
  2. The positive predictive value- the probability that newborns who receive a screen-positive result from the study are actually affected by spinal muscular atrophy - measured by the number of true-positive newborns divided by the combined total of true-positive
To determine the feasibility and reliability of the study screening test and regimen in identifying true negative cases | All outcome measures will be assessed intermittently over the course of the 36 month period of the study
  1. The number of false negative results identified in the Thames Valley and who have actually been screened negative
  2. The specificity value - the ability of the study screening test and regimen to correctly generate a screen-negative result for newborns who are actually not affected by spinal muscular atrophy - measured by the number of true-negative newborns divided by the combined total of true-negative and false-positive newborns (times 100%)
To evaluate the feasibility of performing spinal muscular atrophy screening on newborn dried blood spot with the goal of facilitating early diagnosis of SMA in a UK NBS pathway | All outcome measures will be assessed intermittently over the course of the 36 month period of the study
  The time passed between the birth of newborns to the availability of their SMA screening results
To investigate the epidemiology of spinal muscular atrophy in the Thames Valley | This will be assessed at the end of the 3 year study
  1. The incidence of SMA, measured by the number of diagnostic-positive newborns from the study population divided by the total study population during the study period
  2. The number of SMN2 gene copies and their distribution among diagnostic-positive newborns

OTHER OUTCOMES:
To evaluate whether treatment can be delivered in a timely fashion, consistent with what global SMA screening studies have shown to be able to facilitate | All outcome measures will be assessed intermittently over the course of the 36 month period of the study
  The time passed between the birth of diagnostic-positive newborns to the initiation of their SMA treatment
To evaluate logistic and cost of SMA screening | This will be assessed at the end of the 3 year study
  Human Resources (FTE) and cost associated with NBS

CONTACTS AND LOCATIONS:
Locations (9):
- United Kingdom (9):
  - Buckinghamshire HealthCare Trust, Buckingham
  - Dorset County Hospital (DCHFT), Dorchester
  - Milton Keynes University Hospital NHS Foundation Trust, Milton Keynes
  - University of Oxford UK, Oxford
  - St Mary's Maternity Hospital, Poole
  - Queen Alexandra Hospital, Portsmouth
  - Royal Berkshire NHS Foundation Trust, Reading
  - Salisbury District Hospital, Salisbury
  - Princess Anne Hospital, Southampton

IPD SHARING:
Plan to Share IPD: No